CLINICAL TRIAL: NCT06607588
Title: Selection of Resistant Mutations to Dolutegravir and Associated Drugs in PLWH Treated in Clinical Practice in Chokwé, Mozambique
Brief Title: Selection of Resistant Mutations to Dolutegravir in PLWH Treated in Mozambique
Acronym: REDOCH
Status: Recruiting | Type: Observational
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Other Study IDs: REDOCh study
Record Dates: First submitted 2024-09-17; First posted 2024-09-23 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: HIV; HIV Antiretroviral Therapy (ART) Adherence
Keywords: HIV; ARV; Resistance; DTG; Africa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HIV-1 infected men or women >18 years controlled in the day care center of Chokwé Hospital
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — Not applicable- observational study

SUMMARY:
The HIV infection not fully controlled, despite being under antiretroviral treatment, could make virus resistance against the antiretroviral treatments, making hardest the well control of HIV infection. The purpose of this research study is to confirm or deny if a not fully good controlled HIV infection could develop virus resistance against antiretroviral drugs that can difficult the good control of the HIV infection.

DETAILED DESCRIPTION:
This research study consists of a single visit, in which you will be taken an additional vial of blood to analyze the presence or absence of mutations in your virus to HIV drugs. In addition, other HIV infection routine information will be recorded:

* Demographic data
* HIV infection history data
* Virological failure information
* Laboratory parameters Resistance tests techniques: Genotyping resistance test will be performed from plasma samples in those patients with viral load over 200 copies/ml, using ultracentrifugation if needed (Inzaule, Seth C et al. J Antimicrob Chemother, 2018). Briefly, RNA will be extracted and HIV-1 pol gene will be amplified, followed by a nested-PCR. Amplification products will be purified, quantified and finally diluted and prepared for sequencing following Illumina DNA Sample Preparation Kit protocol (Illumina, San Diego, CA). Samples will finally be pooled and sequenced in a MiSeq System (Illumina). MiSeq sequences will be downloaded from Basespace (Illumina) and analysed using PASeq (IrsiCaixa,Barcelona,ES), v1.4.18 (https://www.paseq.org). The questionnaire about clinical and demographic characteristics will be performed during the study visit

ELIGIBILITY:
Inclusion Criteria:

* Patients able to understand and sign the informed consent form.
* Documented HIV-1 infection.
* Under the first line TLD for at least 6 months.
* At least 3 months follow-up with CV >200c/ml.

Exclusion Criteria:

* Patients <18 years of age.
* Under the first line regime other than TLD.
* Patients with active neoplastic processes.
* Patients with active opportunistic diseases.
* Patients unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1 infected men or women >18 years controlled in the day care center of Chokwé Hospital
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Selection of DRM to dolutegravir and/or tenofovir and/or lamivudine | 3 months
  % of Selection of DRM to dolutegravir and/or tenofovir and/or lamivudine

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Carmelo, Chokwé, Mozambique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Inquérito INSIDA — https://ins.gov.mz/search/INSIDA/(2023)